CLINICAL TRIAL: NCT01319669
Title: Clinical Trial on the Prevention of Thrombocytopenia After First-line Chemotherapy With GC/GP Regimens for Non-small-cell Lung Carcinoma Using Recombinant Human Thrombopoietin (rhTPO)
Brief Title: Clinical Trial on the Prevention of Thrombocytopenia After First-line Chemotherapy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: recruiting too slowly
Sponsor: Chinese Society of Lung Cancer (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Vice President of Guangdong General Hospital, Guangdong Academy of Medical Sciences, Chinese Society of Lung Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-TONG1001
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): rhTPO(recombinant human thrombopoietin) is given on the second, 4th and 9th day of the chemotherapy cycle in a dosage of 15000U once subcutaneously.
  Interventions: Drug: recombinant human thrombopoietin
- Control group (Active Comparator): 15000U of rhTPO(recombinant human thrombopoietin) is given subcutaneously 6 to 24 hours within the end of chemotherapy cycle, that is, the 8th day for 3 consecutive days (d9 to d11)
  Interventions: Drug: recombinant human thrombopoietin

INTERVENTIONS:
Drug: recombinant human thrombopoietin — Recombinant human thrombopoietin injection in 15000U/ml/amp.
  Other Names: rhTPO

SUMMARY:
To assess the efficacy and safety of administration of rhTPO at different time in the treatment of thrombocytopenia caused by first-line GC/GP regimen for non small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This is a randomized, controlled, open-labeled, multicenter clinical trial. The subjects are patients with NSCLC who are going to receive GC/GP regimen chemotherapy.

Vadhan-Raj et al conducted a study in which they administered rhTPO in various ways to patients with sarcoma receiving platinum-containing chemotherapy. The results demonstrated that timing of administration of rhTPO can be adjusted according to the occurrence time of nadir platelet values induced by chemotherapy. The timing of administration of rhTPO in this study was determined based on the above proofs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at the age of 18 to 75 years old
2. Histologically or cytologically diagnosed NSCLC cases
3. Thrombocytopenia occurred in the selected chemotherapy cycle confirmed by double test results with platelet count lower than 75×109/L
4. Fit for chemotherapy (WBC ≥ 4.0×109/L；neutrophil count> 1.5×109/L；PLT ≥ 80×109/L；ALT ≤ 3 times the upper limit of normal range；AST ≤ 3 times the upper limit of normal range；TBil ≤ twice the upper limit of normal range；ECOG PS ≤ 2；without severe cardiopulmonary defects)
5. Expected lifespan over 12 weeks
6. With understanding ability and voluntarily sign informed consent form
7. Be able to comply with the study and follow-up process

Exclusion Criteria:

1. With any unstable systemic diseases including active infection, uncontrolled hypertension, liver diseases, renal diseases or metabolic diseases
2. With uncontrolled brain metastasis symptoms (patients whose brain metastasis controlled over 4 weeks without hormone therapy can still be enrolled)
3. With heart cerebrovascular diseases, congestive heart failure with NYHA above II degree, with unstable angina pectoris, with acute myocardial infarction or cerebral infarction within 6 months
4. Breast-feeding or pregnant women
5. Platelet count over 300×109/L

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
minimum and maximum value of platelet count after chemotherapy | nine weeks
  To evaluate the minimum and maximum value of platelet count after chemotherapy and the value of platelet count and their D-values comparing with the baseline values

SECONDARY OUTCOMES:
The duration when patient's platelet count remains below 50×109/L | nine weeks
  The duration when patient's platelet count remains below 50×109/L, the time (in day) when patient's platelet count increases over 75×109/L and 100×109/L, the amount of platelet infused (number of units of apheresis platelet should be transformed into number of units of platelet concentrate)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, Professor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China